CLINICAL TRIAL: NCT05959057
Title: ERr 731® Formulation Evaluation: A Comparison of Enteric Coated and Micro-coated ERr 731® Formulations
Brief Title: ERr 731® Formulation Evaluation
Acronym: EFE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-002
Record Dates: First submitted 2023-04-24; First posted 2023-07-25 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Menopause
Keywords: Botanical supplement; Formulation; Rhapontic Rhubarb

STUDY DESIGN:
Intervention Model Description: double-blinded, randomized cross-over design in a peri-menopausal/menopausal and preferably symptomatic group of women (target population for commercialization) is best suited to demonstrate equivalent tolerability
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded as to order formulations are received in a standard cross-over design with washout phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteric/Micro Order (Experimental): Subjects will receive randomly two distinct formulations of ERr 731® in a 43 day trial consisting of treatment phase 1 (14-days), washout phase (14-days),treatment phase 2 (14-days): Arm 1 will receive enteric coated ERr 731® during treatment phase 1 and micro-coated ERr 731®during treatment phase 2
  Interventions: Dietary Supplement: ERr 731 - Micro-coated; Dietary Supplement: ERr 731 - Enteric coated
- Micro/Enteric Order (Experimental): Subjects will receive randomly two distinct formulations of ERr 731® in a 43 day trial consisting of treatment phase 1 (14-days), washout phase (14-days),treatment phase 2 (14-days): Arm 2 will receive micro-coated ERr 731® during treatment phase 1 and enteric coated ERr 731®during treatment phase 2
  Interventions: Dietary Supplement: ERr 731 - Micro-coated; Dietary Supplement: ERr 731 - Enteric coated

INTERVENTIONS:
Dietary Supplement: ERr 731 - Micro-coated — natural extract of the Rheum Rhaponticum L plant (Siberian rhubarb). The primary active constituents of ERr 731® are hydroxystilbenes, primarily rhaponticin and desoxyrhaponticin.
Dietary Supplement: ERr 731 - Enteric coated — natural extract of the Rheum Rhaponticum L plant (Siberian rhubarb). The primary active constituents of ERr 731® are hydroxystilbenes, primarily rhaponticin and desoxyrhaponticin.
  Other Names: Estrovera

SUMMARY:
A comparison of an enteric coated and micro-coated formulation of ERr 731®

DETAILED DESCRIPTION:
Current clinical and commercialization experiences have been with enteric-coated formulations of ERr 731®. With the demonstrated safety of this formulation and the absence of anthraquinones in the extract, there is interest in launching a micro-coated, but not enteric-coated, formulation to broaden the commercial availability of ERr 731® in new markets. It is proposed that a double-blinded, randomized cross-over design in a peri-menopausal/menopausal and preferably symptomatic group of women (target population for commercialization) is best suited to demonstrate equivalent tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Ages 35-64, inclusive, preference given to Subjects Ages 45-54, inclusive
* Preference given to symptomatic Subjects; symptoms including vasomotor symptoms, mood disturbances, fatigue, myalgias and arthralgias.

Exclusion Criteria:

* A serious, unstable illness including cardiac, hepatic, renal, gastrointestinal, respiratory, endocrinologic, neurologic, immunologic/rheumatological, or oncological/hematologic disease.
* History of Breast or Uterine cancers.
* Known infection with HIV, Tuberculosis or Hepatitis B or C.
* Hormone Replacement Therapy: All formulations of synthetic estrogens, natural estrogens (estrone, estradiol and estriol) and progestins (including natural progesterone)
* Hormonal Contraceptives: All formulations of synthetic estrogens and progestins
* Botanical Formulations - including phytoestrogens and progesterone-mimetic botanicals (Rhapontic Rhubarb, Soy Phytoestrogens, Hops (8-prenyl naringin) Red Clover, Kudzu, Chaste Tree Berry, Licorice, Resveratrol, Black Cohosh, Dong Quai, etc.)
* Use of Narcotics during the last 30 days
* Use of Anticoagulants during last 30 days
* Use of Corticosteroids during the last 30 days
* Use of controlled substances (other than marijuana or CBD) on a recreational basis during the last 30 days.
* Consumption of more than 3 alcoholic beverages per day (One beverage is a 5-ounce glass of wine, 12 ounces of beer, or one ounce of hard liquor)
* Pregnancy
* Breast Feeding

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Tolerability | 14 days
  Frequency of symptoms of gastrointestinal nature collected on a custom questionnaire

SECONDARY OUTCOMES:
General Tolerability | 14 Days
  Frequency of general symptoms collected on a custom questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Personalized Lifestyle Medicine Center, Gig Harbor, Washington, United States

IPD SHARING:
Plan to Share IPD: No